CLINICAL TRIAL: NCT04106167
Title: Long-term, Non-interventional, Observational Study Following Treatment With Fate Therapeutics FT500 Cellular Immunotherapy
Status: Terminated | Type: Observational
Why Stopped: This study was terminated by the Sponsor.
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: FT-003
Record Dates: First submitted 2019-09-16; First posted 2019-09-26 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Advanced Solid Tumor; Lymphoma; Gastric Cancer; Colorectal Cancer; Head and Neck Cancer; Squamous Cell Carcinoma; EGFR Positive Solid Tumor; HER2-positive Breast Cancer; Hepatocellular Carcinoma; Small-cell Lung Cancer; Renal Cell Carcinoma; Pancreas Cancer; Melanoma; NSCLC; Urothelial Carcinoma; Cervical Cancer; Microsatellite Instability; Merkel Cell Carcinoma
MeSH Terms: conditions — Lymphoma; Stomach Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Carcinoma, Squamous Cell; Carcinoma, Hepatocellular; Small Cell Lung Carcinoma; Carcinoma, Renal Cell; Pancreatic Neoplasms; Melanoma; Carcinoma, Transitional Cell; Uterine Cervical Neoplasms; Microsatellite Instability; Carcinoma, Merkel Cell | interventions — Carboxylesterase

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Treatment with Fate Therapeutics' FT500 Cellular Immunotherapy: Long Term follow-up of subjects who have received an allogeneic, iPSC-derived NK cell in a previous trial.
  Interventions: Genetic: Allogeneic natural killer (NK) cell

INTERVENTIONS:
Genetic: Allogeneic natural killer (NK) cell — No study drug is administered in this study. Subjects who received an allogeneic, iPSC-derived NK cell in a previous trial will be evaluated in this trial for long-term safety and efficacy

SUMMARY:
Subjects who previously took part in the FT500-101 study and received allogeneic NK cell immunotherapy will take part in this long term follow-up study. Subjects will automatically enroll into study FT-003 once they have withdrawn or complete the parent interventional study.

The purpose of this study is to provide long-term safety and survival data for subjects who have participated in the parent study. No additional study drug will be given, but subjects can receive other therapies for their cancer while they are being followed for long term safety in this study.

DETAILED DESCRIPTION:
This is a multicenter, non-interventional, observation study designed to provide long-term safety and efficacy data on subjects who have participated in a prior Fate Therapeutics interventional study of FT500 cellular immunotherapy. Subjects will be contacted every six months (± one month), beginning six months after subject completion or withdrawal from the FT500-101 study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received an allogeneic, iPSC-derived NK cell in a Fate Therapeutics interventional study
* Subjects who have provided Informed consent prior to their study participation

Exclusion Criteria:

* Not Applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with advance solid tumors rolling over from interventional study where they were treated with an allogeneic, iPSC-derived NK cell.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) post-Infusion | From the date of study entry until the date of documented death due to any cause, assessed up to 60 months.
  OS defined as the interval between the date of the first NK cell infusion and the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Fate Trial Disclosure, Study Director — Fate Therapeutics
Locations (4):
- United States (4):
  - UCSD Moores Cancer Center, San Diego, California
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No